CLINICAL TRIAL: NCT07245940
Title: Assessing Safety of Cervical Spine Fusion With NMP® Graft Material: A Retrospective Chart Review
Brief Title: Assessing Safety of Cervical Spine Fusion With NMP®
Status: Not yet recruiting | Type: Observational
Sponsor: Red Rock Regeneration Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-NMP-014
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Spinal Stenosis Cervical
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — N-methylpyrrolidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical Interbody Fusion with NMP: Subject has undergone cervical interbody spine fusion between C2 and T1 where NMP fibers have been used as a bone void filler with minimum of 90-day post-operative follow up data available
  Interventions: Biological: Natural Matrix Protein (NMP) Fibers; Procedure: Cervical interbody fusion

INTERVENTIONS:
Biological: Natural Matrix Protein (NMP) Fibers — Human bone allograft
Procedure: Cervical interbody fusion — Procedure that involves removing the intervertebral disk from the disk space between between 2 or more vertebrae between C2 and T1. When the disk space has been cleared out, the surgeon fills the void between the vertebrae with a bone void filler.

SUMMARY:
The goal of this retrospective chart review study is to assess safety of NMP® in the treatment of cervical spine degenerative conditions by assessing the incidence and nature of AEs in follow-up (minimum of 90 days and up to 2 year post-operatively) as well as reoperation rates.

DETAILED DESCRIPTION:
Interbody fusion is a cornerstone of spinal reconstruction, involving placement of a bone graft within the intervertebral space to achieve fusion between adjacent vertebrae. Autogenous bone graft (ABG), typically harvested from the iliac crest, is considered the gold standard due to its osteogenic potential. However, ABG use is limited by donor site morbidity, infection risk, increased operative time, blood loss, and limited graft availability.

Alternative graft materials, such as recombinant human bone morphogenetic protein-2 (rhBMP-2) and demineralized bone matrix (DBM), have been developed to overcome ABG limitations. While rhBMP-2 is highly osteoinductive, off-label cervical use has been associated with severe complications. DBM offers an osteoconductive scaffold but shows variable clinical performance due to inconsistent BMP content.

Cervical spine fusion is a well-established procedure for cervical spine pathologies, but perioperative complications remain significant. Large population-based studies report overall complication rates of 13-14%, with pulmonary events, postoperative hematomas, and dysphagia among the most common. Advanced age and multiple comorbidities are strong predictors of adverse outcomes, with even a single complication prolonging hospitalization and increasing mortality risk.

Given the limitations of current grafts and the high complication rates of cervical spine fusion surgeries, there is a need to evaluate novel biologically active bone grafts. The NMP® bone graft is designed to promote bone formation and may improve safety and clinical outcomes in cervical fusion.

Accurate assessment of adverse events is critical; this study will use the validated SAVES-V2 system to standardize complication reporting, capture severity, and quantify the clinical and economic impact of cervical spine fusion surgery-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated with NMP® for Cervical (C2-T1) Interbody fusion (2022-2025) at the study site.
2. Minimum of 90-day post-operative follow up data available

Exclusion Criteria:

* Patients with no follow-up data within 3 months from the surgery date due to missed postoperative appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include up to 300 patients who have been treated with Induce Biologics NMP™ during cervical interbody fusion. All subjects who meet all inclusion criteria and do not meet any exclusion criteria will be included in the study. It is expected that enrollment will take 4-5 months to complete.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event Reporting | 90 days - 24 months postoperatively
  assessment of the incidence and nature of AEs. Complications determined to be related to NMP® within at least 3 months post-op will be collected and reported as part of the primary outcome of this study.
Re-operation Rates | 90 days - 24 months postoperatively
  Re-operation rates determined to be related to NMP® within at least 3 months post-op will be collected and reported as part of the primary outcome of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Alabama Back Institute, Jasper, Alabama, United States

IPD SHARING:
Plan to Share IPD: No